CLINICAL TRIAL: NCT01585428
Title: A Phase II Study of Lymphodepletion Followed by Autologous Tumor-Infiltrating Lymphocytes and High-Dose Aldesleukin for Human Papillomavirus-Associated Cancers
Brief Title: Immunotherapy Using Tumor Infiltrating Lymphocytes for Patients With Metastatic Human Papillomavirus-Associated Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120116; 12-C-0116
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Cervical Cancer; Oropharyngeal Cancer; Vaginal Cancer; Anal Cancer; Penile Cancer
Keywords: Immunotherapy; HPV-Associated Cancers; Cervical Cancer; Oropharyngeal Cancer; HPV Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Oropharyngeal Neoplasms; Vaginal Neoplasms; Anus Neoplasms; Penile Neoplasms; Papillomavirus Infections | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cervical (Experimental): Patients will receive a non-myeloablative lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous (IV) infusion of Young tumor infiltrating lymphocytes (TIL) plus high dose IV aldesleukin.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Young TIL; Drug: Aldesleukin
- NonCervical (Experimental): Patients will receive a non-myeloablative lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous (IV) infusion of Young tumor infiltrating lymphocytes (TIL) plus high dose IV aldesleukin
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Young TIL; Drug: Aldesleukin

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 25 mg/m(2)/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml in 5% dextrose in water (D5W) over 1 hr.
  Other Names: Cytoxan
Biological: Young TIL — Cells will be infused intravenously (i.v.) on the Patient Care Unit over 20 to 30 minutes (between one and four days after the last dose of fludarabine).
  Other Names: TIL
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
  Other Names: Proleukin

SUMMARY:
Background:

The human papillomavirus (HPV) can cause a number of cancers, including cervical and throat cancers. The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy that involves taking white blood cells from patients' tumors, growing them in the laboratory in large numbers, and then giving the cells back to the patient. These cells are called Tumor Infiltrating Lymphocytes, or TIL and we have given this type of treatment to over 200 patients with melanoma. Researchers want to know if TIL shrink s tumors in people with human papilloma virus (HPV)-related cancer. In this study, we are selecting a specific subset of white blood cells from the tumor that we think are the most effective in fighting tumors and will use only these cells in making the tumor fighting cells.

Objective:

The purpose of this study is to see if these specifically selected tumor fighting cells can cause HPV-related cancers to shrink and to see if this treatment is safe.

Eligibility:

- Adults age 18-66 with HPV-related cancer who have a tumor that can be safely removed.

Design:

Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed.

Surgery: If the patients meet all of the requirements for the study they will undergo surgery to remove a tumor that can be used to grow the TIL product.

Leukapheresis: Patients may undergo leukapheresis to obtain additional white blood cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}

Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the TIL cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.

Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits will take up to 2 days.

DETAILED DESCRIPTION:
Background:

* Metastatic or locally advanced refractory/recurrent human papillomavirus (HPV)-associated malignancies (cervical, vulvar, vaginal, penile, anal, and oropharyngeal) are incurable and poorly palliated by standard therapies.
* Administration of autologous tumor infiltrating lymphocytes (TIL) generated from resected metastatic melanoma can induce objective long-term tumor responses.
* Young TIL can be generated from HPV-associated tumors.

Objectives:

* To determine if autologous Young TIL infused in conjunction with high dose aldesleukin following a non-myeloablative lymphodepleting preparative regimen can mediate tumor regression in patients with metastatic or locally advanced refractory/recurrent HPV-associated cancer.
* To study immunologic correlates associated with Young TIL therapy for HPV-associated cancers.
* To determine the toxicity of this treatment regimen.

Eligibility:

- Patients greater than or equal to 18 years old with a pathologically confirmed diagnosis of metastatic or locally advanced refractory/recurrent HIPV-16+ or HPV-18+ human papillomavirus-associated cancer.

Design:

* Patients will undergo biopsy or resection to obtain tumor for generation of autologous TIL cultures and autologous cancer cell lines.
* All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day intravenous (IV)) on days -7 and -6 and fludarabine (25 mg/m(2)/day IV) on days -5 through -1.
* On day 0 patients will receive between 1 times 10 (9) to 2 times 10(11) young TIL and then begin high dose aldesleukin (720,000 IU/kg IV every 8 hours for up to 15 doses).
* Clinical and immunologic response will be evaluated about 4-6 weeks after TIL infusion.
* Initially, 18 evaluable patients will be enrolled in two cohorts; patients with cervical cancer and those with non- cervical cancer. For each cohort, if 0 to 2 of the 18 patients experience a clinical response, then no further patients will be enrolled. If 3 or more of the first 18 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 35 evaluable patients have been enrolled in each cohort. Up to 73 patients may be enrolled over approximately 3-4 years.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable metastatic or locally advanced refractory/recurrent malignancies that are human papilloma virus 16 (HPV-16) or human papilloma virus 18 (HPV-18) high HPV positive by in situ hybridization (ISH) or polymerase chain reaction (PCR) or any cancer from the uterine cervix..
2. All patients must have received at least one standard chemotherapy or chemoradiotherapy.
3. Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible.
4. Greater than or equal to 18 years of age and less than or equal to age 70.
5. Able to understand and sign the Informed Consent Document
6. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
7. Life expectancy of greater than three months
8. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
9. Serology:

   * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
   * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcription - polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
10. Women of child bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
11. Hematology

    * Absolute neutrophil count greater than 1000/mm(3) without the support of filgrastim
    * White blood cell (WBC) greater than or equal to 3000/mm(3)
    * Platelet count greater than or equal too 100,000/mm(3)
    * Hemoglobin greater than 8.0 g/dl
12. Chemistry:

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to to 2.5 times the upper limit of normal
    * Serum creatinine less than or equal to to 1.6 mg/dl
    * Total bilirubin less that or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
13. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

    Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria in Section 2.1.1.
14. More than four weeks must have elapsed since any prior radiation therapy.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy treatment on the fetus or infant.
2. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Concurrent systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of coronary revascularization or ischemic symptoms.
8. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%.
9. Documented LVEF of less than or equal to 45% tested in patients with i) clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or ii) age greater than or equal 60 years old.
10. Active Bleeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-04-13 (Actual); Primary Completion 2016-04-09 (Actual); Study Completion 2016-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaturvedi AK, Engels EA, Pfeiffer RM, Hernandez BY, Xiao W, Kim E, Jiang B, Goodman MT, Sibug-Saber M, Cozen W, Liu L, Lynch CF, Wentzensen N, Jordan RC, Altekruse S, Anderson WF, Rosenberg PS, Gillison ML. Human papillomavirus and rising oropharyngeal cancer incidence in the United States. J Clin Oncol. 2011 Nov 10;29(32):4294-301. doi: 10.1200/JCO.2011.36.4596. Epub 2011 Oct 3. PMID 21969503
- [Background] Rosenberg SA, Yang JC, Sherry RM, Kammula US, Hughes MS, Phan GQ, Citrin DE, Restifo NP, Robbins PF, Wunderlich JR, Morton KE, Laurencot CM, Steinberg SM, White DE, Dudley ME. Durable complete responses in heavily pretreated patients with metastatic melanoma using T-cell transfer immunotherapy. Clin Cancer Res. 2011 Jul 1;17(13):4550-7. doi: 10.1158/1078-0432.CCR-11-0116. Epub 2011 Apr 15. PMID 21498393
- [Background] Ryerson AB, Peters ES, Coughlin SS, Chen VW, Gillison ML, Reichman ME, Wu X, Chaturvedi AK, Kawaoka K. Burden of potentially human papillomavirus-associated cancers of the oropharynx and oral cavity in the US, 1998-2003. Cancer. 2008 Nov 15;113(10 Suppl):2901-9. doi: 10.1002/cncr.23745. PMID 18980273
- [Result] Stevanovic S, Draper LM, Langhan MM, Campbell TE, Kwong ML, Wunderlich JR, Dudley ME, Yang JC, Sherry RM, Kammula US, Restifo NP, Rosenberg SA, Hinrichs CS. Complete regression of metastatic cervical cancer after treatment with human papillomavirus-targeted tumor-infiltrating T cells. J Clin Oncol. 2015 May 10;33(14):1543-50. doi: 10.1200/JCO.2014.58.9093. Epub 2015 Mar 30. PMID 25823737
- [Derived] Malekzadeh P, Pasetto A, Robbins PF, Parkhurst MR, Paria BC, Jia L, Gartner JJ, Hill V, Yu Z, Restifo NP, Sachs A, Tran E, Lo W, Somerville RP, Rosenberg SA, Deniger DC. Neoantigen screening identifies broad TP53 mutant immunogenicity in patients with epithelial cancers. J Clin Invest. 2019 Mar 1;129(3):1109-1114. doi: 10.1172/JCI123791. Epub 2019 Feb 4. No abstract available. PMID 30714987
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0116.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervical | NonCervical
Started | 18 | 11
Completed | 17 | 11
Not Completed | 1 | 0
Not completed — Death during treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical | NonCervical | Total
Number analyzed (Participants) | 18 | 11 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 11 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (11.4) | 54.9 (4.5) | 47.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 6 | 24
  Male | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 11 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 11 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Objective Clinical Response
Description: Patients must have a partial response (PR) or complete response (CR) at least 4 months after cell infusion to count towards clinical response. Clinical response is assessed by the Response Criteria in Solid Tumors (RECIST) v1.0. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Complete response is disappearance of all target lesions. Progression is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum LD.
Time Frame: 4 months after cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical | NonCervical
Number analyzed (Participants) | 18 | 11
Participants
  Partial Response | 3 | 2
  Complete Response | 2 | 0
  Progressive Disease | 12 | 8
  Stable Disease | 1 | 1

2. Secondary Outcome: Number of Patients With Serious and Non-serious Adverse Events
Description: Here is the number of serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0). A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. A non-serious adverse event is any untoward medical occurrence.
Time Frame: 51 months and 18 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical | NonCervical
Number analyzed (Participants) | 18 | 11
Participants | 18 | 11

ADVERSE EVENTS:
Time Frame: 51 months and 18 days
Arm/Group | Cervical | NonCervical
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/11
Serious Adverse Events (participants affected / at risk) | 4/18 | 2/11
Other Adverse Events (participants affected / at risk) | 17/18 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervical (N=18) | NonCervical (N=11)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Death not associated with CTCAE term: Disease progression NOS (General disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 2 (2) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 1 (1) | 2 (2) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 0 (0) — (ANC <1.0 x 10e) ::Blood
Infection (Infections and infestations) | 1 (1) | 0 (0) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Oral cavity-gums (gingivitis)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Obstruction, GU::Ureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervical (N=18) | NonCervical (N=11)
Hemoglobin (Blood and lymphatic system disorders) | 16 (16) | 8 (8)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 10 (10) | 8 (8)
Lymphopenia (Blood and lymphatic system disorders) | 17 (18) | 10 (10)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 17 (17) | 11 (11)
Platelets (Blood and lymphatic system disorders) | 17 (17) | 11 (11)
Hypotension (Cardiac disorders) | 2 (2) | 3 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hemorrhage, GI:: Lower GI NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 6 (6) | 3 (3) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection (Infections and infestations) | 6 (6) | 6 (6) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 2 (2) | 2 (2)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 2 (2) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0)
Pain::Abdomen NOS (General disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Oliguria) (Renal and urinary disorders) | 2 (2) | 0 (0)
Rigors/chills (General disorders) | 0 (0) | 1 (1)
Incontinence, anal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mental status (Nervous system disorders) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GU::Vagina (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) | 0 (0) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Upper airway NOS
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 1 (1) — (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 0 (0) | 1 (1)
Pain::Back (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Obstruction, GU::Ureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain::Head/Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-07-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT01585428/ICF_000.pdf
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT01585428/Prot_001.pdf